CLINICAL TRIAL: NCT06808750
Title: Schistosoma Haematobium Diagnostic Test Performance in the Elimination Setting Pemba, Tanzania
Brief Title: Performance of Tests for Schistosoma Haematobium Diagnosis
Acronym: SchistoBreak-D
Status: Completed | Type: Observational
Sponsor: Stefanie Knopp (Other)
Collaborators: Public Health Laboratory Ivo de Carneri (Other); Enaiblers AB (Industry); Erasmus Medical Center (Other); Leiden University Medical Center (Other); Natural History Museum, United Kingdom (Other Government)
Responsible Party: Sponsor-Investigator, Stefanie Knopp, Principal Investigator, Swiss Tropical & Public Health Institute
Organization: Swiss Tropical & Public Health Institute (Other)
Other Study IDs: 1687; PR00P3_179753 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2025-01-08; First posted 2025-02-05 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Schistosoma Haematobium
Keywords: schistosomiasis; diagnosis; elimination; control
MeSH Terms: conditions — Schistosomiasis haematobia; Schistosomiasis; Disease | interventions — Microscopy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The microscope slides containing the urine filters will be stored for quality control for approximately 6-12 months and disposed after quality control at PHL-IdC.
  The left overs of any collected urine sample from participants of the diagnostic accuracy study on Day 1-5 will be stored in 50 ml plastic tubes labelled with the participant ID code in a freezer at PHL-IdC at -20°C for further use for research purposes.
  The DNA extracted from fresh and frozen urine samples for RPA, PeakPCR and qPCR will be labelled with the participant ID code, stored at +4°C and shipped to LUMC for examination with qPCR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants of initial screening: Schoolchildren that attend classes in grades 3-6 in each of the two study schools will be invited to submit one urine sample that will be tested with a single urine filtration (Day 1).
  Interventions: Diagnostic Test: S. haematobium egg detection by single urine filtration; Diagnostic Test: Haematuria assessment using reagent strips
- Participants of diagnostic study: All schoolchildren that are tested S. haematobium-positive children in the initial screening plus a sex-adjusted random selection of initially negative-screened children will be included in the diagnostic study. These children will be invited to submit five urine samples in total, over five days (Day 1-5). All samples (Day 1-5) will be tested with a single urine filtration. Samples collected on Day 5 will be tested with all investigated diagnostic tests.
  Interventions: Diagnostic Test: S. haematobium egg detection by single urine filtration; Diagnostic Test: S. haematobium egg detection by quintuple urine filtration; Diagnostic Test: S. haematobium egg detection by artificial intelligence (AI) microscopy; Diagnostic Test: Haematuria assessment using reagent strips; Diagnostic Test: S. haematobium antigen detection by up-converting reporter particle-lateral flow circulating anodic antigen assay (UCP-LF CAA); Diagnostic Test: S. haematobium DNA detection by recombinase polymerase amplification assay (RPA); Diagnostic Test: S. haematobium DNA detection by qPCR

INTERVENTIONS:
Diagnostic Test: S. haematobium egg detection by single urine filtration — The urine samples of children participating in the initial screening will be tested with a single urine filtration by human microscopy.
Diagnostic Test: S. haematobium egg detection by quintuple urine filtration — Five urine samples will be collected from children participating in the diagnostic study over five days. Each of the five urine samples collected per participant will be tested with a single urine filtration by human microscopy.
  Groups: Participants of diagnostic study
Diagnostic Test: S. haematobium egg detection by artificial intelligence (AI) microscopy — The urine samples collected on Day 5 of the diagnostic study will be tested with artificial intelligence (AI) microscopy.
  Groups: Participants of diagnostic study
Diagnostic Test: Haematuria assessment using reagent strips — The urine samples collected from children participating in the initial screening and in the diagnostic study, respectively, will be tested with reagent strips.
Diagnostic Test: S. haematobium antigen detection by up-converting reporter particle-lateral flow circulating anodic antigen assay (UCP-LF CAA) — The urine samples collected on Day 5 of the diagnostic study will be tested with the up-converting reporter particle-lateral flow circulating anodic antigen assay (UCP-LF CAA).
  Groups: Participants of diagnostic study
Diagnostic Test: S. haematobium DNA detection by recombinase polymerase amplification assay (RPA) — The urine samples collected on Day 5 of the diagnostic study will be tested with the recombinase polymerase amplification assay (RPA).
  Groups: Participants of diagnostic study
Diagnostic Test: S. haematobium DNA detection by qPCR — The urine samples collected on Day 5 of the diagnostic study will be tested with qPCR
  Groups: Participants of diagnostic study

SUMMARY:
Urogenital schistosomiasis caused by infection with the blood fluke Schistosoma haematobium is a debilitating disease. The World Health Organization (WHO) has set the goal to eliminate schistosomiasis as a public health problem globally by 2030 and to interrupt transmission in selected areas. Many years of control interventions and mass drug administration have reduced substantially the prevalence and infection intensities in several areas. In areas with an infection prevalence <10%, the WHO suggests to continue population preventive chemotherapy with praziquantel at the same or reduced frequency, or to use a clinical approach of test-and-treat. In areas that have achieved interruption of transmission, elimination needs to be validated and post-elimination surveillance be implemented.

For determination of infection prevalence thresholds, for test-and-treat, for validation of elimination and for pre- and post-elimination surveillance, reliable diagnostic tools are needed.

In a single-centre study conducted in Pemba, United Republic of Tanzania, the investigators aim to assess the accuracy and performance of standard and new diagnostic tests for S. haematobium diagnosis for use in elimination settings.

The primary objective of the study is to assess the sensitivity and specificity of all investigated diagnostic tests, using the S. haematobium egg count results of five urine filtrations conducted on five urine samples collected over five consecutive days as reference test.

Secondary objectives are:

* To assess the sensitivity and specificity of all investigated diagnostic tests, using latent class analyses.
* To assess the sensitivity and specificity of all investigated diagnostic tests, in relation to S. haematobium infection intensity, calculated as mean egg count derived from the egg counts in five urine samples collected over 5 consecutive days.
* To assess the sensitivity and specificity of all investigated diagnostic tests, in relation to S. haematobium infection intensity, calculated from the egg counts of the urine sample that was analysed with the respective test and urine filtration.
* To assess the sensitivity and specificity of all investigated diagnostic tests, using the results of the up-converting reporter particle-lateral flow circulating anodic antigen assay (UCP-LF CAA) as reference test.
* To assess the sensitivity and specificity of all investigated molecular diagnostic tests, using the results of the qPCR as reference test.
* To assess the cost and time needed for the implementation of single or multiple-throughput tests.

Our study will evaluate the accuracy and performance of diagnostic tests, in a formerly highly endemic setting that is now approaching elimination (Pemba), and will hence provide important information about which tests can be recommended for threshold determination, and test-and-treat and surveillance.

ELIGIBILITY:
Inclusion Criteria:

Subjects fulfilling all of the following inclusion criteria are eligible for the initial screening:

* Attendance of grade 3, 4, 5, or 6 in study school
* Randomized to participate in initial screening
* Written informed consent signed by the parents
* Written assent signed by the participant if aged12-17 years old

Subjects fulfilling all of the following inclusion criteria are eligible for the diagnostic study:

* Attendance of grade 3, 4, 5, or 6 in study school
* Randomized to participate in initial screening
* Written informed consent signed by the parents
* Written assent signed by the participant if aged12-17 years old
* S. haematobium-positive urine filtration result in initial screening OR
* S. haematobium-negative urine filtration result in initial screening, but randomized for participation in diagnostic study

Exclusion Criteria:

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject in the initial screening:

* Not attending any study school
* Not attending grade 3, 4, 5 or 6
* Not randomized to participate in initial screening
* No written informed consent signed by the parents submitted
* No written assent signed by the participant if aged12-17 years old submitted
* S. haematobium-negative urine filtration result in initial screening, and not randomized for participation in diagnostic performance study
* Clinical significant sever disease

The presence of any one of the following exclusion criteria will lead to the exclusion of the subject in the diagnostic study:

* Not attending any study school
* Not attending grade 3, 4, 5 or 6
* Not randomized to participate in initial screening
* No written informed consent signed by the parents submitted
* No written assent signed by the participant if aged12-17 years old submitted
* S. haematobium-negative urine filtration result in initial screening, and not randomized for participation in diagnostic performance study
* Clinical significant sever disease

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children from Pemba Island, United Republic of Tanzania, that attend one among the two pre-selected study primary schools in grade 3, 4, 5 or 6.
Sampling Method: Probability Sample
Enrollment: 801 (Actual)
Dates: Start 2025-02-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Accuracy of tests for S. haematobium diagnosis when compared with a single urine filtration | From enrollment to the end of the study after 6 weeks
  The primary endpoint will be the sensitivity of the investigated diagnostic tests to detect S. haematobium related markers by the examination of a single sample.
  The primary outcome variable will be the number of S. haematobium infected individuals detected through each test.

SECONDARY OUTCOMES:
Sensitivity of each diagnostic test (human microscopy, AI microscopy, reagent strips, RPA, UCP-CAA, qPCR). | From enrollment to the end of the study after 6 weeks
  Sensitivity is defined as the proportion of positive test results out of all truly positive samples. Reference tests are human microscopy, UCP-CAA, qPCR or a combination thereof, performed with the same urine sample (human microscopy, UCP-CAA, qPCR) or quintuple urine samples (human microscopy).

OTHER OUTCOMES:
Specificity of each diagnostic test (human microscopy, AI microscopy, reagent strips, RPA, UCP-CAA, qPCR). | From enrollment to the end of the study after 6 weeks.
  Specificity is defined as the proportion of negative test results out of all truly negative samples. Reference tests are human microscopy, UCP-CAA, qPCR or a combination thereof, performed with the same urine sample (human microscopy, UCP-CAA, qPCR) or quintuple urine samples (human microscopy).
Correlation of infection markers. | From enrollment to the end of the study after 6 weeks.
  Correlation of the amount of infection markers measured by each test (human microscopy: number of S. haematobium eggs, AI microscopy: number of S. haematobium eggs, reagent strips: microhaematuria grading, RPA: fluorescence level, UCP-CAA: amount of CAA antigen, qPCR: cycle-threshold values).
Costs of each diagnostic test (human microscopy, AI microscopy, reagent strips, RPA, UCP-CAA, qPCR). | 6 month, from start of orders of equipment and material to end of laboratory work.
  Costs are defined as the financial costs incurred by each test for equipment, consumables, and staff time to perform the test.
Time to conduct each diagnostic test (human microscopy, AI microscopy, reagent strips, RPA, UCP-CAA, qPCR). | From enrollment to the end of the study after 6 weeks.
  Amount of time spent completing each test.

CONTACTS AND LOCATIONS:
Overall Officials: Stefanie Knopp, PhD, Principal Investigator — Swiss Tropical & Public Health Institute; Said M Ali, MSc, Study Director — Public Health Laboratory Ivo de Carneri
Locations (1):
- Public Health Laboratory - Ivo de Carneri (PHL-IdC), Chake Chake, Pemba Island, Tanzania

IPD SHARING:
Plan to Share IPD: Yes
* There are data transfer agreements (DTAs) in place between the Public Health Laboratory-Ivo de Carneri (PHL-IdC) in Pemba and the Swiss Tropical and Public Health Institute (Swiss TPH), Switzerland; Leiden University Medical Centre (LUMC), The Netherlands; Natural History Museum (NHM), London, UK; and Enaiblers, Sweden.
  * Anonymized data will be curated and stored for an unlimited period in the data repository "Infectious Diseases Data Observatory" (IDDO; https://www.iddo.org/) and/or Zenodo (https://zenodo.org/).
  * Data may be shared with other researchers upon request.